CLINICAL TRIAL: NCT05308888
Title: Impact of Local Tissue Inflammation on Intramyocardial Conduction Pathways Post Percutaneous Valve : Evaluation by Positron Emission Tomography on Exploratory Cohort
Acronym: IMPACT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC21.0255 (IMPACT)
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All patients will have to undergo an 18F-FDG PET-CT.
  Interventions: Diagnostic Test: 18F-FDG PET-CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET-CT — The 18F-FDG PET-CT will be performed in the nuclear medicine department of the CHU of Brest. For this exam, the administration of 2-3 MBq/kg of 18F-FDG ([18F]F-fluorodeoxyglucose) will be performed to the patient in a single intravenous injection.

SUMMARY:
Aortic valve stenosis is the most common valve disease leading to surgical or percutaneous intervention in Europe and North America. Percutaneous aortic valve replacement (TAVI) is currently recommended for the management of patients with symptomatic aortic stenosis and with high; very high operative risk of aortic valve replacement surgery or intermediate operative risk of aortic valve replacement surgery after a benefit-risk assessment by a heart team and operative contraindication to conventional aortic valve replacement surgery. These indications are supported by the 2017 European Cardiology guidelines.

This technique of percutaneous arterial valve implantation is most often performed via the femoral route, under local anesthesia, with placement of a prosthetic biological valve in the aortic position, impacting it into the patient's native aortic valve.

TAVI has been shown to be superior to medical treatment in patients with a aortic valve stenosis at very high operative risk of conventional aortic valve replacement surgery. However, the occurrence of atrioventricular conduction disorders (de novo left bundle branch block (LBBB) or complete AVB) remains the most frequent complication after TAVI. Therefore, the rate of pacemaker (PM) implantation after TAVI remains high, ranging from 2% to 51%, with an average rate of 13%.

Pacemaker implantation has several deleterious effects (increased hospitalization time, desynchronization of the left ventricle by permanent right ventricular pacing, exposure of the patient to procedural complications of pacemaker placement, and possible increase in the final cost to society of the initial hospitalization.

Not all patients who received a pacemaker post TAVI implantation use their PM. The rate of Pacemaker dependency and therefore of patients who actually use their pacemaker is approximately 33-36% at 1 year after percutaneous valve implantation.

In view of all the potentially deleterious consequences of post TAVI pacemaker implantation, it is therefore necessary to know which patients really justify pacemaker implantation after percutaneous valve implantation.

The purpose of this study is to investigate diagnostic imaging criteria that may be predictive of the occurrence of intramyocardial conduction disorders post TAVI implantation. Although some patients present only transient conductive disturbances, the impact of tissue inflammation of the intramyocardial conduction pathways after TAVI remains to be understood.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (>18 years of age);
* Patient with aortic stenosis defined by aortic valve area ≤ 1cm2 (or indexed aortic valve area ≤ 0.6 cm2/m2 body surface area), OR transvalvular peak velocity ≥ 4 m/s OR transvalvular mean gradient ≥ 40 mmHg, as assessed by transthoracic echocardiography performed in a patient at rest;
* Symptomatic patient with: dyspnea ≥ New-York Heart Association (NYHA) stage 2 OR pathological stress test with onset of symptoms on exertion, blood pressure drop, or rhythm disorder on exertion OR Asymptomatic with Left Ventricular Ejection Fraction < 50% ;
* Patient with vascular anatomy compatible with percutaneous femoral valve implantation;
* Patient affiliated to or benefiting from a health insurance plan;
* Patient who has provided free, informed and written consent.

Exclusion Criteria:

* Patient with a pacemaker or triple chamber defibrillator prior to TAVI implantation;
* Patient with a uni or bicuspid aortic valve;
* Patient with severe left ventricular dysfunction LVEF < 30%;
* Patient with other significant valve disease : aortic insufficiency ≥ grade 3, mitral insufficiency ≥ grade 3 or tight mitral stenosis ;
* Patient with iliofemoral vascular anatomy preventing safe passage of the valve;
* Patient with a pre-existing bioprosthesis or mechanical prosthesis at TAVI in any position;
* Inability or refusal to consent;
* Pregnant or breastfeeding woman;
* Patient under judicial protection or family habilitation;
* Patient deprived of liberty by judicial or administrative decision, under guardianship or curatorship;
* Patient with life expectancy < 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a conductive disorder | Up to 5 days after TAVI's implantation
  The primary end point is "occurrence of conductive disturbance": 1) complete BAV, 2) high-grade BAV, 3) LBBB, 4) RBBB, 5) BAV1; assessed by the performance of post-percutaneous valve implantation electrocardiograms (ECGs) during the initial patient's hospitalization.

SECONDARY OUTCOMES:
Number of participants requiring pacemaker implantation | Up to 5 days after TAVI's implantation, 1, 6 and 12 months
  Number of participants requiring pacemaker implantation post-TAVI
Simulation rate of pacemaker | 1 and 6 month
  Simulation rate of the right ventricular lead of the pacemaker at 1 and 6 months after TAVI's implantation
Occurrence of a conductive disorder | 6 month
  Occurrence of a conductive disorder (atrioventricular blocks or high-grade atrioventricular block or left buncle branch block or right bundle branch block or atrioventricular block grade 1) within 6 months of discharge from TAVI's hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient.
Access Criteria: Data access requests will be reviewed by the internal committee of BrestUH. Requestors will be required to sign and complete a data access agreement.